CLINICAL TRIAL: NCT02802085
Title: A Prospective Observational 5 Year Follow-up on a Historical Consecutive Cohort of 100 Primary Total Knee Arthroplasty (TKA) Cases Treated With the Posterior-stabilized VEGA System® PS
Brief Title: VEGA Prospective Kiel
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Frictionless GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: AAG-I-H-1319
Record Dates: First submitted 2016-05-25; First posted 2016-06-16 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Degenerative Osteoarthritis; Rheumatoid Arthritis
Keywords: Total Knee Arthroplasty; Total Knee Replacement; TKA; TKR; Stiffness of Knee; Deformity; Knee Joint; Instability; Post-traumatic; Arthrosis
MeSH Terms: conditions — Joint Diseases; Arthritis, Rheumatoid; Congenital Abnormalities; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee Arthroplasty: Vega Knee Arthroplasty
  Interventions: Device: VEGA Knee

INTERVENTIONS:
Device: VEGA Knee — TKA

SUMMARY:
Voluntary Post-Marketing Clinical Follow-up (PMCF) as part of the post marketing surveillance plan for the product under investigation.

For this PMCF only CE-marked medical devices have been used and will be used within their intended purpose and no additional invasive or other stressful examinations have been or are to be carried out (acc. to MPG §23b).

DETAILED DESCRIPTION:
This non-interventional clinical study (NIS) is conducted to clinically confirm the safety and performance of the Aesculap® VEGA System® PS components under routine conditions. The VEGA System® PS is an established TKA design, and there is a long-lasting experience in the use of PS components in particular; thus a NIS is thought to be sufficient to give the required confirmation. For this NIS only CE-marked medical devices have been used and will be used within their intended purpose and no additional invasive or other stressful examinations have been and are to be carried out (acc. to MPG §23b). This voluntary NIS is part of the post-marketing surveillance for the product under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received primary TKA at the study site five to six years ago using the product under investigation because of the following severe knee joint conditions that could not be treated through other therapies:
* degenerative osteoarthritis,
* rheumatoid arthritis,
* posttraumatic arthritis,
* symptomatic knee instability, knee stiffness or deformation of the knee joint
* Age at the time of surgery ≥ 18 years
* Patient signed informed consent

Exclusion Criteria:

* Age younger than 18 years at the time of surgery
* Any prior joint replacement at the index knee
* Patient did not sign informed consent
* All cases not listed under indications (according to IfU)
* All cases showing any contraindication (according to IfU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Revision (non-survival) rate | 5 years
  The objective of the study is to collect clinical 5 year outcome information on the product under investigation when used in routine clinical practice.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 5 years
  Changes of the total Knee injury and Osteoarthritis Outcome Score (KOOS) from the preoperative baseline to the 5 year postoperative assessment
Physical Component Summary (PCS-12) of SF-12® Health Survey (SF-12) | 5 years
  Changes of the total SF-12® Health Survey (SF-12) from the preoperative baseline to the 5 year postoperative assessment
Mental Component Summary (MCS-12) of SF-12® Health Survey (SF-12) | 5 years
  Changes of the total SF-12® Health Survey (SF-12) from the preoperative baseline to the 5 year postoperative assessment
Pain | 5 years
  Changes of anterior knee pain according to the Waters and Bentley rating system from the preoperative baseline to the 5 year postoperative assessment
Knee Score (KS) of Knee Society Score (KSS) | 5 years
  The Knee Score (KS) of the Knee Society Score (KSS) at the 5 year postoperative assessment
Functional Score (FS) of Knee Society Score (KSS) | 5 years
  The Functional Score (FS) of the Knee Society Score (KSS) at the 5 year postoperative assessment

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Gerdesmeyer, Professor, Principal Investigator — orthopedics
Locations (1):
- MEDBALTIC GmbH c/o Mare Klinikum, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerdesmeyer L, Glowalla C, Lasic I, Al Muderis M, Weuster M, Klueter T. The Vega advanced third generation posterior stabilized total knee arthroplasty system enables the restoration of range of motion for high demanding daily activities - A 5-years follow-up study. PLoS One. 2024 May 13;19(5):e0302885. doi: 10.1371/journal.pone.0302885. eCollection 2024. PMID 38739584